CLINICAL TRIAL: NCT03006185
Title: Pretreatment With Ablative Fractional Laser and Microdermabrasion Before Photodynamic Therapy for Actinic Keratoses in Field-cancerized Skin
Brief Title: Laser and Microdermabrasion Before Photodynamic Therapy for Actinic Keratoses in Field-cancerized Skin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Principal Investigator, Merete Haedersdal, Professor and Senior Physician, Bispebjerg Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: H-16023991; 2015-002331-18 (EudraCT Number)
Record Dates: First submitted 2016-12-09; First posted 2016-12-30 (Estimated); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Actinic Keratosis; Sun Damaged Skin; Solar Keratosis; Solar Skin Damage
MeSH Terms: conditions — Keratosis, Actinic | interventions — Lasers

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion (Experimental): WIthin each participant, two 50 cm2 adjacent test areas were randomized to laser or microdermabrasion pretreatment prior to daylight photodynamic therapy.
  Interventions: Device: Ablative Fractional Carbon Dioxide (CO2) Laser; Device: Microdermabrasion

INTERVENTIONS:
Device: Ablative Fractional Carbon Dioxide (CO2) Laser — One 50 cm2 test area was randomized to pretreatment using a fractional 2940 nm Er:YAG laser (Joule®; Sciton Inc., Palo Alto, CA, USA). To remove hyperkeratosis, a fully-ablative 4 mm handpiece was optionally applied, followed by a single pass of a fractional Profrax 430 handpiece for all AKs. Subsequent field treatment consisted of a single pass of the Profrax 430 handpiece over the entire test area. Immediately after pretreatment, a 0.5 mm layer of methyl aminolevulinate (Metvix ® cream 16%; Galderma, Paris, France) was applied. After 30 minutes, patients were exposed to 2 hours of ambient daylight, according to approved procedure. After light exposure, cream was wiped off and test areas were covered for the remainder of the day.
Device: Microdermabrasion — Another adjacent 50 cm2 test area was exposed to microdermabrasion using an MD pad with 58.5 µm-diameter particles (Ambu® Skin Prep Pads 2121M; Ambu A/S, Ballerup, Denmark). Lesion-directed treatment consisted of an increasing number of swipes concentrated to AK lesions. During field treatment, multiple swipes were applied in perpendicular directions over the entire test area. Immediately after pretreatment, a 0.5 mm layer of methyl aminolevulinate (Metvix ® cream 16%; Galderma, Paris, France) was applied. After 30 minutes, patients were exposed to 2 hours of ambient daylight, according to approved procedure. After light exposure, cream was wiped off and test areas were covered for the remainder of the day.

SUMMARY:
Comparison of treatment efficacy and safety of pretreatment with ablative fractional laser versus microdermabrasion combined with large-area photodynamic therapy with methyl aminolevulinate for actinic keratoses

DETAILED DESCRIPTION:
For each study participant, two test areas (A and B) are demarcated in the same anatomical region, with each area containing no less than 5 actinic keratoses (AKs). Test areas are randomized to receive skin pretreatment of EITHER ablative fractional laser OR microdermabrasion prior to photodynamic therapy using methyl aminolevulinate.

Efficacy, local skin reactions and safety of both test areas are evaluated over a 12-15 week follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with two skin areas of at least 50 cm2 with a minimum of 5 actinic keratoses (AKs) grade I-III, chronically sun damaged "field" changes in one of the following anatomical regions: face, scalp, upper chest.
* Patients who have given written informed consent and are believed to be capable of following the study protocol.
* Fertile women must have a negative pregnancy test (urine-hCG) at the time of inclusion and use anti-contraception (oral contraceptives, intrauterine device, gestagen depot injection, subdermal implantation, vaginal ring, transdermal depot bandage or sterilisation) during the study.

Exclusion Criteria:

* Patients that have within the last month received local treatment in the test areas.
* Pregnant or nursing patients.
* Patients with porphyria
* Patients with skin cancer, keratoacanthoma, or other infiltrating tumors within the test areas.
* Patients with a tendency to develop hypertrophic scars or keloids.
* Patients with a known allergy to Metvix cream
* Patients that are believe unlikely to follow the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08; Primary Completion 2016-11 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merete Haedersdal, MD, Dr. Med, Principal Investigator — Bispebjerg Hospital

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Test areas
Groups:
- Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion: Intra-individual design. "All study participants" are grouped into a single arm. Two adjacent skin areas (test areas) on each participant was allocated through randomization to two different interventions: 1) Pretreatment with Ablative Fractional (AFL) CO2 laser OR 2) Microdermabrasion (MD) prior to standard daylight photodynamic therapy.
  Description of intervention: Ablative Fractional CO2 laser: CO2 laser treatment is randomly allocated to one of two tests areas within each study participant. Laser treatment consists of targeted ablation of actinic keratoses and field laser treatment of the entire test area. After laser treatment, application of methyl aminolevulinate (MAL), a topical photosensitizing agent, is performed. The test area thereafter undergoes 2 hours of daylight photodynamic therapy.
  Microdermabrasion: Microdermabrasion (processing of the skin with a sandpaper-like material) is randomly allocated to one of two tests areas in each study participant. Microdermabrasion treatment consists of targeted treatment of actinic keratoses and field treatment of the entire test area. Afterwards, application of methyl aminolevulinate (MAL), a topical photosensitizing agent, is performed. The test area then undergoes 2 hours of daylight photodynamic therapy.
Period: Overall Study
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Started | 18; 36 Test areas (Since all participants had two test areas each, all participants received both interventions (18 test areas received CO2 and 18 test areas received microdermabrasion))
Number of Test Areas Recieving AFL | 18; 36 Test areas
Number of Test Areas Receiving MD | 18; 36 Test areas
Completed | 18; 36 Test areas
Not Completed | 0; 0 Test areas

BASELINE CHARACTERISTICS:
Population: Each participant had two skin areas that individually were randomized to receive either microdermabrasion or ablative fractional laser prior to photodynamic therapy. Thus, with 18 participants, we had 36 test areas.
Units Other Than Participants: Skin areas
Groups:
- Split Person Design: Pretreatment With Ablative Fractional Carbon Dioxide Laser or Microdermabrasion: Two 50 cm2 test areas (Test Area A and B) are demarcated on the skin of each study participant. One test area is randomized to receive the intervention: Ablative Fractional Carbon Dioxide (CO2) Laser prior to standard daylight photodynamic therapy. The other test area is randomized to receive the intervention: microdermabrasion prior to standard daylight photodynamic therapy.
  Ablative Fractional Carbon Dioxide (CO2) Laser: Ablative Fractional Carbon Dioxide (CO2) Laser treatment is randomly allocated to one of two tests areas in each study participant. Laser treatment consists of targeted ablation of actinic keratoses and field laser treatment of the entire test area. After laser treatment, application of methyl aminolevulinate (MAL), a topical photosensitising agent, is performed. The test area thereafter undergoes 2 hours of daylight photodynamic therapy.
  Microdermabrasion: Microdermabrasion (processing of the skin with a sandpaper-like material) is randomly allocated to one of two tests areas in each study participant. Microdermabrasion treatment consists of targeted treatment of actinic keratoses and field treatment of the entire test area. Afterwards, application of methyl aminolevulinate (MAL), a topical photosensitising agent, is performed. The test area then undergoes 2 hours of daylight photodynamic therapy.
Arm/Group | Split Person Design: Pretreatment With Ablative Fractional Carbon Dioxide Laser or Microdermabrasion
Number analyzed (Participants) | 18
Number analyzed (Skin areas) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 15
Age, Continuous [Mean (Full Range); unit: years] | 72.5 [52 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 12
Region of Enrollment [Number; unit: participants]
  Denmark | 18

OUTCOME MEASURES:

1. Primary Outcome: Complete Clearance (%) of Actinic Keratoses (AKs)
Description: Percentage clearance of baseline actinic keratoses (AKs), determined by the ratio of AK lesions that are clinically resolved 12-15 weeks after treatment compared to the AK number at baseline.
Time Frame: 12-15 weeks post-treatment
Population: Percentage AK clearance in test areas receiving either AFL (18) or microdermabrasion (18) assisted daylight PDT treatment
Measure: Mean (Full Range); unit: percentage (%) of AK clearance
Units Other Than Participants: Test areas
Groups:
- Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion: Intra-individual design of 18 participants. "All study participants" are grouped into a single arm. Two adjacent skin areas (test areas) on each participant is allocated through randomization to two different interventions: 1) Pretreatment with Ablative Fractional (AFL) CO2 laser OR 2) Microdermabrasion (MD) prior to standard daylight photodynamic therapy. Thus, each participants received both inventions (18 test areas received AFL and 18 test areas received MD).
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
Number analyzed (Test areas) | 36
percentage (%) of AK clearance
  Ablative Fractional Laser | 81 [53 to 100]
  Microdermabrasion | 60 [24 to 94]

2. Secondary Outcome: New Actinic Keratoses (AKs)
Description: Number of new actinic keratoses (AKs) identified clinically 12-15 weeks after treatment and that were not present at the baseline evaluation.
Time Frame: 12-15 weeks post-treatment
Measure: Median (Inter-Quartile Range); unit: New AK lesions
Units Other Than Participants: Test areas
Groups:
- Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion: Intra-individual design of 18 participants. "All study participants" are grouped into a single arm. Two adjacent skin areas (test areas) on each participant is allocated through randomization to two different interventions: 1) Pretreatment with Ablative Fractional (AFL) CO2 laser OR 2) Microdermabrasion (MD) prior to standard daylight photodynamic therapy. Thus, each participants receives both inventions (18 test areas received AFL and 18 test areas received MD).
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
Number analyzed (Test areas) | 36
New AK lesions
  Ablative Fractional Laser | 0 [0 to 0.25]
  Microdermabrasion | 1 [0 to 2]

3. Secondary Outcome: Severity of Local Skin Reactions (LSRs)
Description: Local skin reactions scale (min:0; better and max: 3; worse) used to grade each of the following parameters: erythema, edema, crusting, pustules, ulceration and scabbing, scaling.
  The severity of each evaluated clinically on a 4-point scale where 0 = none, 1= mild, 2= moderate and 3= severe.
  With 7 parameters the sum of all scores will produce a maximum composite score of 21.
Time Frame: Day 3-6 post treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Test areas
Groups:
- Pretreatment: Two 50 cm2 test areas (Test Area A and B) are demarcated on the skin of each study participant. One test area is randomized to receive the intervention: Ablative Fractional Carbon Dioxide (CO2) Laser prior to standard daylight photodynamic therapy. The other test area is randomized to receive the intervention: microdermabrasion prior to standard daylight photodynamic therapy.
  Ablative Fractional Carbon Dioxide (CO2) Laser: Ablative Fractional Carbon Dioxide (CO2) Laser treatment is randomly allocated to one of two tests areas in each study participant. Laser treatment consists of targeted ablation of actinic keratoses and field laser treatment of the entire test area. After laser treatment, application of methyl aminolevulinate (MAL), a topical photosensitizing agent, is performed. The test area thereafter undergoes 2 hours of daylight photodynamic therapy.
Arm/Group | Pretreatment
Number analyzed (Participants) | 18
Number analyzed (Test areas) | 36
score on a scale
  Ablative Frational Laser | 7 [5 to 10]
  Microdermabrasion | 4 [2 to 6]

4. Secondary Outcome: Degree of Sun Damage
Description: Sun damage is evaluated clinically on a 4 point scale where 0 = none, 1= mild, 2= moderate and 3= severe sun damage.
Time Frame: 12-15 weeks post-treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Skin Areas
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
Number analyzed (Skin Areas) | 36
score on a scale
  Ablative Fractional Laser | 1 [0 to 2]
  Microdermabrasion | 2 [1 to 2.25]

5. Secondary Outcome: Treatment-related Pain
Description: Patient-reported pain during treatments is evaluated using the visual analog scale (VAS) where 0= no pain and 10= worst imaginable pain.
Time Frame: during treatment (day 0)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
units on a scale
  Ablative Fractional Laser | 3 [2 to 4]
  Microdermabrasion | 5 [4 to 6]

6. Secondary Outcome: Treatment-related Side Effects
Description: Side effects are evaluated over the course 12-15 weeks following treatment. In addition to unforeseen adverse events, specific side effects including the clinical presence of infection, scarring, hypopigmentation and hyperpigmentation are recorded.
Time Frame: up to 12-15 weeks post-treatment
Measure: Number; unit: Local Staf infection
Units Other Than Participants: Test areas
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
Number analyzed (Test areas) | 36
Local Staf infection
  Ablative Fractional Laser | 3
  Microdermabrasion | 1

7. Secondary Outcome: Investigator-reported Cosmesis (Clinical Evaluation)
Description: Cosmetic appearance of treated areas is evaluated by investigators clinically (scores on a scale) using a 4-point scale where 0 = none, 1= acceptable, 2= good and 3= excellent outcome.
Time Frame: 12-15 weeks post-treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Test areas
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
Number analyzed (Test areas) | 36
score on a scale
  Ablative Fractional Laser | 3 [2 to 3]
  Microdermabrasion | 2 [1.5 to 2]

8. Secondary Outcome: Patient-reported Cosmesis
Description: Cosmetic appearance is evaluated by patients at the end of the study (scores on a scale) using a 4 point scale where 0 = none, 1= acceptable, 2= good and 3= excellent
Time Frame: 12-15 weeks post-treatment
Measure: Median (Inter-Quartile Range); unit: score on a scale
Units Other Than Participants: Test areas
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
Number analyzed (Test areas) | 36
score on a scale
  Ablative Fractional Laser | 3 [2 to 3]
  Microdermabrasion | 2 [1 to 2]

9. Secondary Outcome: Patient Pretreatment Preference
Description: Patients were asked to report which pretreatment they preferred: Laser, microdermabrasion, or no preference
Time Frame: 12-15 weeks post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Split-Person Design: Ablative Fractional Carbon Dioxide (CO2) Laser vs Microdermabrasion
Number analyzed (Participants) | 18
Participants
  Ablative Fractional Laser | 12
  Microdermabrasion | 4
  No Preference | 2

ADVERSE EVENTS:
Groups:
- Split-Person: Ablative Fractional Carbon Dioxide Laser or Microdermabrasion: Intra-individual design of 18 participants. "All study participants" are grouped into a single arm. Two adjacent skin areas (test areas) on each participant is allocated through randomization to two different interventions: 1) Pretreatment with Ablative Fractional (AFL) CO2 laser OR 2) Microdermabrasion (MD) prior to standard daylight photodynamic therapy. Thus, each participants receives both inventions (18 test areas received AFL and 18 test areas received MD).
Arm/Group | Split-Person: Ablative Fractional Carbon Dioxide Laser or Microdermabrasion
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 3/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Split-Person: Ablative Fractional Carbon Dioxide Laser or Microdermabrasion (N=18)
Infection in test areas treated with AFL (Infections and infestations) | 3 (3) — Staph aureus infection was noted in 3/18 test areas pretreated with ablative fractional laser
Infection in test areas treated with MD (Infections and infestations) | 1 (1) — Staph aureus infection was noted in 1/18 test areas pretreated with microdermabrasion

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes